CLINICAL TRIAL: NCT01472679
Title: Body Composition: a Predictor of Mortality in Subjects Over 65 Years
Status: Completed | Type: Observational
Sponsor: Genton Graf Laurence (Other)
Responsible Party: Sponsor-Investigator, Genton Graf Laurence, Principal investigator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: 11-161R
Record Dates: First submitted 2011-11-07; First posted 2011-11-16 (Estimated); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: External Causes of Morbidity and Mortality
Keywords: fat mass; fat free mass; body mass index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate whether body composition is associated with a higher risk of mortality in subjects ≥ 65 years.

DETAILED DESCRIPTION:
Study centre: University Hospitals of Geneva Study type: retrospective study Study duration (anticipated): 1 year for collection of data(1.10.2011-1.12.2012)and 3 months for statistical analysis and writing, leading to the completion of the study by march 2013 Study hypothesis: A low fat-free mass (FFM) and a high fat mass (FM) are associated with a higher risk of mortality in subjects ≥ 65 years.

Aims: The primary objective is to evaluate the relationship between body composition and mortality in men and women ≥ 65 years, while taking into account co-morbidities. The secondary objectives are to compare this relationship a) with the relationship of body mass index (BMI) and mortality, b) with the relationship of body composition changes and mortality, c) between healthy subjects and subgroups of patients with chronic diseases Methods: Included are all subjects who had a measurement of body composition by bioelectrical impedance analyses, performed in the HUG from 1990 until december 2011. Excluded are subjects living abroad. Body composition measurements will be retrieved from DPI and 4D which preceded the use of DPI in nutrition and is presently only used for research. Diseases and specific laboratory values at time of body composition measurement will be retrieved simultaneously. Mortality will be retrieved from the population registers for death.

Statistics: The relationship between body composition and mortality, in the total population and subgroups of patients with chronic diseases, will be evaluated by Cox regression, adjusted for age, gender and co-morbidities. The variance of mortality (adjusted R2) related to FFM will be compared to that related to BMI and FFM loss.

ELIGIBILITY:
Inclusion Criteria:

* All subjects ≥ 65 years included in previous studies on body composition by bioelectrical impedance analysis performed in the Nutrition Unit since 1990 until December 2011.
* All patients ≥ 65 years who had a measurement of body composition by bioelectrical impedance analysis performed in clinical routine by the Nutrition Unit and the dietitians of the University Hospital of Geneva since 1990 until December 2011, while hospitalized or not.

Exclusion Criteria:

* Subjects living in another country than Switzerland at time of body composition measurement

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: This is a historical cohort study of prospectively collected measurements of body composition performed by bioelectrical impedance analysis, between 1990 and 2011.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Actual)
Dates: Start 2016-10; Primary Completion 2018-05 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Mortality | Mortality from 1 January 1990 to 31 December 2011
  Report if the subject died or not until 31st December 2011

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Genton, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- University Hospital, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Graf CE, Herrmann FR, Genton L. Relation of Disease with Standardized Phase Angle among Older Patients. J Nutr Health Aging. 2018;22(5):601-607. doi: 10.1007/s12603-018-1034-4. PMID 29717760
- [Derived] Graf CE, Karsegard VL, Spoerri A, Makhlouf AM, Ho S, Herrmann FR, Genton L. Body composition and all-cause mortality in subjects older than 65 y. Am J Clin Nutr. 2015 Apr;101(4):760-7. doi: 10.3945/ajcn.114.102566. Epub 2015 Feb 11. PMID 25833973